CLINICAL TRIAL: NCT02225574
Title: An Open-Label, Phase I/II Study of Nilotinib (Tasigna) and MEK-162 (ARRY-162) Used in Combination for Patients With Refractory or Advanced Chronic Myeloid Leukemia and Philadelphia Positive Acute Leukemia (Protocol CAMN107AUS41T)
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Slow Accrual - Only 1 patient enrolled in Phase 1 - Study never went to Phase II
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: Array BioPharma (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2014-0128; NCI-2015-00044 (Registry Identifier: NCI CTRP)
Record Dates: First submitted 2014-08-22; First posted 2014-08-26 (Estimated); Last update posted 2020-02-12 (Actual); Status verified 2020-02

CONDITIONS: Leukemia
Keywords: Leukemia; Advanced phase chronic myeloid leukemia; refractory chronic phase chronic myeloid leukemia; CML; Accelerated phase; (AP); Blast phase; (BP); Philadelphia-positive acute leukemia; MEK-162; Nilotinib; AMN107; Tasigna; Questionnaires; Surveys
MeSH Terms: conditions — Leukemia; Leukemia, Myeloid, Chronic-Phase; Blast Crisis | interventions — binimetinib; nilotinib; Surveys and Questionnaires

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Advanced CML + Philadelphia positive Acute Leukemia-Group 1 (Experimental): Phase 1 Starting dose of MEK-162: 30 mg by mouth twice a day of a 28 day cycle.
  Phase 1 Starting dose of Nilotinib: 400 mg by mouth twice a day of a 28 day cycle.
  Questionnaires completed and the end of cycle 1, 2, 3, 6, 9, and 12.
  Phase 2 Starting dose of MEK-162: MTD from Phase 1 to be taken by mouth twice a day starting on Day 1 of a 28 day cycle.
  Phase 2 Starting dose of Nilotinib: MTD from Phase 1 to be taken by mouth twice a day starting on Day 2 of a 28 day cycle.
  Interventions: Drug: MEK-162; Drug: Nilotinib; Behavioral: Questionnaires
- Chronic Phase CML - Group 2 (Experimental): Phase 1 Starting dose of MEK-162: 30 mg by mouth twice a day of a 28 day cycle.
  Phase 1 Starting dose of Nilotinib: 400 mg by mouth twice a day of a 28 day cycle.
  Questionnaires completed and the end of cycle 1, 2, 3, 6, 9, and 12.
  Phase 2 Starting Dose of Nilotinib: MTD from Phase 1 by mouth twice a day starting on Day 1 of a 28 day cycle.
  Phase 2 Starting Dose of MEK-162: MTD from Phase 1 by mouth twice a day starting on Day 8 of a 28 day cycle.
  Interventions: Drug: MEK-162; Drug: Nilotinib; Behavioral: Questionnaires

INTERVENTIONS:
Drug: MEK-162 — Phase 1: Advanced CML + Philadelphia positive Acute Leukemia-Group 1 Starting Dose of MEK-162: 30 mg by mouth twice a day on starting on Day 1 of a 28 day cycle.
  Phase 2 Advanced CML + Philadelphia positive Acute Leukemia-Group 1 Starting dose of MEK-162: MTD from Phase 1 to be taken by mouth twice a day starting on on Day 1 of a 28 day cycle.
  Phase 1 Chronic Phase CML - Group 2 Starting dose of MEK-162: 30 mg by mouth twice a day of a 28 day cycle.
  Phase 2 Chronic Phase CML - Group 2 Starting Dose of MEK-162: MTD from Phase 1 by mouth twice a day starting on Day 8 of a 28 day cycle.
Drug: Nilotinib — Phase 1 Advanced CML + Philadelphia positive Acute Leukemia-Group 1 Starting Dose of Nilotinib: 400 mg by mouth twice a day of a 28 day cycle.
  Phase 2 Advanced CML + Philadelphia positive Acute Leukemia-Group 1 Starting dose of Nilotinib: MTD from Phase 1 to be taken by mouth twice a day starting on Day 2 of a 28 day cycle.
  Phase 1 Chronic Phase CML - Group 2 Starting dose of Nilotinib: 400 mg by mouth twice a day of a 28 day cycle.
  Phase 2 Chronic Phase CML - Group 2 Starting Dose of Nilotinib: MTD from Phase 1 by mouth twice a day starting on Day 1 of a 28 day cycle.
  Other Names: AMN107; Tasigna
Behavioral: Questionnaires — Questionnaires completed and the end of cycle 1, 2, 3, 6, 9, and 12.
  Other Names: Surveys

SUMMARY:
The goal of this clinical research study is to find the highest tolerated dose of the combination of nilotinib and MEK-162 that can be given to patients with CML or acute leukemia. Researchers also want to learn if the drug combination can help to control the disease. The safety of the drug combination will also be studied.

DETAILED DESCRIPTION:
Study Groups:

If you are found to be eligible to take part in this study, you will be assigned to a study group based on when you join this study. Up to 5 groups of up to 6 participants will be enrolled in Phase 1 of the study, and up to 60 participants will be enrolled in Phase 2.

If you are enrolled in Phase 1, the dose of nilotinib and MEK-162 you receive will depend on when you joined this study. The first group of participants will receive the starting dose combination level. The next group will receive a higher dose of MEK-162 than Group 1, if no intolerable side effects were seen. If intolerable side effects are seen, the next group may receive a lower dose level of nilotinib and/or MEK-162. This will continue until the highest tolerable combination dose is found.

If you are enrolled in Phase 2, you will receive nilotinib and MEK-162 at the highest dose that was tolerated in Phase 1.

Study Treatment:

You will take nilotinib and MEK-162 two times every day by mouth.

Participants enrolled in Phase 1 of the study will start taking MEK-162 on Day 1 and nilotinib on Day 2.

Participants in Phase 2 of the study will be divided in 2 groups: one group will start MEK-162 on Day 1 and nilotinib on Day 2, while the other group will start MEK-162 on Day 1 and nilotinib on Day 8. You will be placed in a Phase 2 treatment group based on the characteristics of your disease type.

You will be given a drug diary and asked to write down what time you take the study drugs every day. Bring in any unused study drugs and bottles to each study visit.

Each cycle is 28 days.

If the disease does not appear to get better after 1 or 3 cycles, you may be able to receive a higher dose of the study drug as long as you are not already receiving the highest dose planned for this study. The study doctor will tell you if you can receive a higher dose.

Study Visits:

On Days 1 and 8 of Cycle 1:

* You will have a physical exam.
* Blood (about 2-3 tablespoons) and urine will be collected for routine tests.
* You will have an EKG.

At the end of Cycle 1:

* You will have a physical exam.
* Blood (about 2-3 tablespoons) and urine will be collected for routine tests.
* You will have an EKG and either a MUGA scan or an ECHO.
* You will complete a questionnaire about how you are feeling.
* If the doctor thinks it is needed, you will have a bone marrow aspirate to check the status of the disease.

At the end of Cycles 2, 3, and every 3 cycles after that (6, 9, 12, and so on):

* You will have a physical exam.
* Blood (about 2-3 tablespoons) and urine will be collected for routine tests.
* You will have an EKG.
* You will complete a questionnaire about how you are feeling.

At the end of Cycles 2, 3, 6, 9, and 12, blood (about 3-4 tablespoons each time) will be drawn for tests to check how the disease is responding to therapy. If the doctor thinks it is needed, these tests may be performed more often.

Every 8-12 weeks, you will have a MUGA scan or an ECHO.

You will have an eye exam by an eye doctor at the end of Cycles 2, 3, 6, 9, and 12, and then every 3 months after that until the End of Study Visit.

You will have blood draws and/or bone marrow aspirations at any time that the doctor thinks it is needed while you are on study.

Length of Study:

You can take up to 12 cycles of nilotinib and MEK-162 on study. If the disease responds a certain way (called a hematological response) while you are on study, you may be able to continue taking the study drugs longer than 12 months, as long as the doctor thinks you are benefiting from the treatment. Even if the disease has not responded in this way, you may be able to continue taking the study drugs if the doctor thinks it is in your best interest. You will no longer be able to take the study drug if the disease gets worse, if intolerable side effects occur, or if you are unable to follow study directions.

Your participation on the study will be over after the follow-up visits.

End-of-Study Visit:

If you come off study before the end of Cycle 12, the following tests and procedures will be performed:

* You will have a physical exam.
* Blood (about 2-3 tablespoons) and urine will be collected for routine tests.
* You will have an EKG and either an ECHO or a MUGA scan.
* You will have an eye exam by an eye doctor.
* You will complete a questionnaire about how you are feeling.
* If the doctor thinks it is needed, you will have a bone marrow aspirate to check the status of the disease.

If you come off study at the end of Cycle 12, you will not have the End of Study visit.

Follow-Up:

You will be called about 30 days after you go off study and asked if you have had any side effects and/or any new treatment(s). This call will last about 5 minutes.

This is an investigational study. Nilotinib is FDA approved and commercially available to treat CML and philadelphia-positive acute leukemia. MEK-162 is not FDA approved or commercially available. It is currently being used for research purposes only. The combination of nilotinib and MEK-162 to treat CML and Philadelphia-positive acute leukemia is investigational. The study doctor can explain how the study drugs are designed to work.

Up to 90 patients will take part in this study. All will be enrolled at MD Anderson Cancer Center.

ELIGIBILITY:
Inclusion Criteria:

1. Patients 18 years of age or older with advanced CML (CML-AP, CML-BP and Philadelphia chromosome-positive acute leukemia) or refractory chronic phase CML are eligible, as defined as follows: The phase I portion of the study will be conducted first in advanced phase (accelerated phase CML, blast phase CML or Philadelphia-positive acute leukemia) patients. Once MTD is identified, a cohort of 6 patients with CML chronic phase who have failed prior therapy with at least two tyrosine kinase inhibitor will be treated at the MTD to determine if this dose is also acceptable for chronic phase patients. The phase II will be conducted in two treatment arms as follows: Treatment Arm A (Advanced phase disease) and treatment Arm B (Therapy for CP-CML refractory/resistant/suboptimally responding to at least two prior TKI's)
2. (Cont - Inclusion Criteria #1) CML-AP is defined by the presence of one of the following: a. 15-29% blasts in peripheral blood (PB) or bone marrow (BM), b.>20% basophils in PB or BM, c.>30% blasts plus promyelocytes (with blasts <30%) in PB or BM, d.<100 x109/L platelets unrelated to therapy, or Clonal cytogenetics evolution (i.e., the presence of cytogenetic abnormalities other than the Philadelphia chromosome) except if only present at the time of diagnosis and not associated with other features of accelerated phase. CML-BP is defined by the presence of >/=30% blasts in the bone marrow and/or peripheral blood or the presence of extramedullary disease, with myeloid or lymphoid blast morphology. Philadelphia-chromosome acute leukemias are eligible and defined by >/=20% blasts in the peripheral blood or bone marrow at the time of diagnosis.
3. Patients with advanced phase CML or acute leukemia must have failed at least one prior TKI. Patients with chronic phase CML must have failed, have resistance or suboptimal response to at least two tyrosine kinase inhibitors, or have intolerance to two prior tyrosine kinase inhibitors. For patient with prior intolerance, they should have received at least 2 TKI and experienced intolerance to one TKI and resistance/suboptimal
4. (Cont - Inclusion Criteria #3) a. Failure to tyrosine kinase inhibitors will be defined per European-Leukemia-Net (ELN) recommendations b.Resistance or suboptimal response to at least two prior Abl-kinase inhibitor, specifically: i.Chronic-phase with resistance to imatinib, dasatinib, nilotinib, bosutinib or ponatinib defined as 1. Loss of CCyR at any time or failure to achieve CCyR after >/=18 months 2. Loss of MCyR at any time or failure to achieve PCyR after >/=12 months 3. Failure to achieve any CyR (ie, >/= 65% Ph+) after >/= 6 months 4. Hematologic relapse or failure to achieve CHR after >/=3 months ii. Chronic-phase with suboptimal response to imatinib, defined as 1. Failure to achieve PCyR after >/= 6 months 2. Failure to achieve CCyR after >/=12 months iii. Chronic-phase with suboptimal response to nilotinib, bosutinib, dasatinib or ponatinib, defined as 1. Failure to achieve PCyR after >/= 3 months 2. Failure to achieve CCyR after >/= 6 months of therapy
5. Patients with cytogenetic BCR-Abl variants and additional chromosomal abnormalities ('clonal evolution') will be eligible. Cytogenetics to be performed, but results are not required to start therapy in patients with hematologic progression
6. Patients who have failed nilotinib, including those who are refractory to nilotinib at any dose or have relapsed on nilotinib at any dose will be eligible for the study. Patients currently on nilotinib will continue on their prescribed dose of nilotinib and MEK-162 will be added based on the current cohort level in phase I or at the established MTD in phase II. In the instance the nilotinib dose is greater than the current cohort (in phase 1) or the MTD (in phase 2) patients will be dose reduced to the dosage as prescribed by protocol and then dose escalated as allowed in protocol at the PIs discretion.
7. For the phase I portion of the study, patients who had received prior therapy with nilotinib should have been able to tolerate the dose equivalent to the starting dose of nilotinib in the dose level at which the patient is being entered. Patients who previously received nilotinib but never at the dose being proposed are eligible provided they tolerated the maximum dose they were prescribed with no grade 3 or 4 toxicity not responding to optimal management.
8. Patients must have been off all prior therapy for CML for 2 weeks prior to start of study therapy and recovered from the toxic effects of that therapy. Exceptions to these are hydroxyurea and TKIs (including but not limited to imatinib, nilotinib, dasatinib, ponatinib and bosutinib), which should be discontinued ≥48 hrs prior to the start of therapy. Patients who are receiving nilotinib prior to enrollment do not have to discontinue this agent prior to start of study therapy
9. Eastern Cooperative Oncology Group (ECOG) performance status </=2
10. Men and women of childbearing potential should practice effective methods of contraception. Men and women of childbearing potential are defined as: a male that has not been surgically sterilized or female that has not been amenorrheic for at least 12 consecutive months or that has not been surgically sterilized. Patients must use birth control during the study and for 3 months after the last dose of study drug if they are sexually active.
11. Adequate organ function: Serum creatinine </=2.0 mg/dl or creatinine clearance >/=60 mL/min, Direct bilirubin </=2.0xULN (unless considered due to leukemia involvement), Alanine aminotransferase (ALT) </=2.5xULN (</=5.0xULN if considered due to leukemic involvement.)
12. Adequate cardiac function: left ventricular ejection fraction (LVEF) >/= 50% as determined by a multigated acquisition (MUGA) scan or echocardiogram, QTc interval </= 480 ms;
13. Women of childbearing potential must have a pregnancy test at screening.
14. Signed informed consent.

Exclusion Criteria:

1. Impaired cardiac function including any one of the following: a. Inability to monitor the QT interval on ECG b. Congenital long QT syndrome or a known family history of long QT syndrome. c. Clinically significant resting brachycardia (<45 beats per minute) d. QTc > 480 msec on baseline ECG. If QTc >450 msec and electrolytes are not within normal ranges, electrolytes should be corrected and then the patient re-screened for QTc e. Impaired cardiovascular function or clinically significant cardiovascular diseases, including any of the following: History of acute coronary syndromes (including myocardial infarction, unstable angina, coronary artery bypass grafting, coronary angioplasty, or stenting) <6 months prior to screening, Symptomatic chronic heart failure, history or current evidence of clinically significant cardiac arrhythmia and/or conduction abnormality <6 months prior to screening except atrial fibrillation and paroxysmal supraventricular tachycardia
2. History of Gilbert's syndrome.
3. Uncontrolled arterial hypertension despite medical treatment
4. Prior therapy with a MEK- inhibitor
5. History or current evidence of retinal vein occlusion (RVO) or current risk factors for RVO (e.g. uncontrolled glaucoma or ocular hypertension, history of hyperviscosity or hypercoagulability syndromes)
6. History of retinal degenerative disease;
7. Patients with washout period < 6 weeks from the last dose of ipilimumab or other immunotherapy
8. Known positive serology for HIV, active hepatitis B, and/or active hepatitis C infection
9. Patients who have neuromuscular disorders that are associated with elevated CK (e.g., inflammatory myopathies, muscular dystrophy, amyotrophic lateral sclerosis, spinal muscular atrophy)
10. Patients who are planning on embarking on a new strenuous exercise regimen after first dose of study treatment. Muscular activities, such as strenuous exercise, that can result in significant increases in plasma CK levels should be avoided while on MEK162 treatment
11. Patients currently receiving treatment with strong CYP3A4 inhibitors who cannot discontinue such treatment or be switched to a different medication prior to starting study drug are excluded from study entry. Strong CYP3A4 inhibitors include the following medications: itraconazole, ketoconazole, miconazole, voriconazole; amprenavir, atazanavir, fosamprenavir, indinavir, nelfinavir, ritonavir; ciprofloxacin, clarithromycin, diclofenac, doxycycline, enoxacin, isoniazid, ketamine, nefazodone, nicardipine, propofol, quinidine, telithromycin.
12. Patients receiving treatment with any medications that have the potential to prolong the QT interval who cannot discontinue such treatment or be switched to a different medication prior to starting study drug are excluded from the study entry. A list of anti-arrhythmic drugs and other drugs that may prolong the QT interval is added in protocol section 8.5 (page 53).
13. Impaired gastrointestinal (GI) function or active GI disease that may significantly alter the absorption of study drug in the opinion of the treating physician (e.g., active ulcerative diseases, uncontrolled nausea, uncontrolled vomiting, uncontrolled diarrhea, active malabsorption syndrome, small bowel resection within last 1 year or gastric bypass surgery within last 1 year).
14. Another active primary malignant disease, which requires systemic treatment (chemotherapy or radiation)
15. History of significant congenital or acquired bleeding disorder unrelated to cancer
16. Major surgery within 4 weeks prior to Day 1 of the study or who have not recovered from prior surgery.
17. Pregnant or nursing (lactating) women, where pregnancy is defined as the state of a female after conception and until the termination of gestation, confirmed by a positive human chorionic gonadotropin (hCG) laboratory test
18. Women of child-bearing potential, defined as all women physiologically capable of becoming pregnant, unless they are using highly effective methods of contraception throughout the study and for 3 months after study drug discontinuation. Highly effective methods of contraception are further defined.
19. Patients who are eligible, willing and able to receive an allogeneic stem cell transplant within 6 weeks are not eligible.
20. Sexually active males unless they use a condom during intercourse while taking the drug and for 3 months after stopping treatment and should not father a child in this period. A condom is required to be used also by vasectomized men in order to prevent delivery of the drug via seminal fluid;
21. History of non-compliance to medical regimens or inability to grant consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2015-03-11 (Actual); Primary Completion 2017-02-02 (Actual); Study Completion 2017-02-02 (Actual)

PRIMARY OUTCOMES:
Maximum Tolerated Dose (MTD) of MEK-162 and Nilotinib | 28 days
  MTD defined as maximum daily oral dose at which <33% of patients experience a dose limiting toxicity (DLT) during first 28 days. DLT defined by events that are clinically significant and at least possibly related to study drug occurring during the first 4 weeks of therapy. Toxicities reported on a scale of 1-4 according to the NCI criteria Common Terminology Criteria for Adverse Events (CTCAE).

SECONDARY OUTCOMES:
Response Rate for Advanced CML and Philadelphia-Positive Acute Leukemia | 28 days
  For CML response defined as major hematological response (MaHR) at the end of the 1st cycle. For Philadelphia-positive acute leukemia response defined as achievement of complete remission(CR)/CR with incomplete platelet recovery (CRp)/ CR with insufficient hematological recovery (CRi)/partial remission (PR)/morphologic leukemia free (MLF) at the end of the 1st cycle.
  For Philadelphia-positive acute leukemia response defined as improvement in one response category (eg, from complete hematological response [CHR] to any cytogenetic response, from minor cytogenetic response to partial cytogenetic response, from partial cytogenetic response to complete cytogenetic response, from complete cytogenetic response to major molecular response [MMR]) at end of the 3rd cycle.
Response Rate for Chronic Phase CML | After 3, 28 day cycles
  Response defined as improvement in one response category (eg, from complete hematological response [CHR] to any cytogenetic response, from minor cytogenetic response to partial cytogenetic response, from partial cytogenetic response to complete cytogenetic response, from complete cytogenetic response to major molecular response [MMR]) at end of the 3rd cycle.

CONTACTS AND LOCATIONS:
Overall Officials: Naval Daver, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- University of Texas MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org